CLINICAL TRIAL: NCT04741997
Title: A Randomized Pilot Trial of Adjuvant Therapy Based on Pathologic Response After Neoadjuvant Encorafenib and Binimetinib in Advanced Melanoma
Brief Title: Adjuvant Therapy Based on Pathologic Response After Neoadjuvant Encorafenib Binimetinib in Melanoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20641
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Melanoma Stage III; Melanoma Stage IV; BRAF V600 Mutation
Keywords: Skin
MeSH Terms: conditions — Melanoma | interventions — encorafenib; binimetinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Surveillance (Active Comparator): Participants will receive 24 weeks of neoadjuvant encorafenib and binimetinib and then proceed to planned resection. If participants have pathologic complete response they will receive adjuvant treatment for 24 weeks. Imaging will be conducted every 12 weeks for at least one year after surgery, and every 24 weeks for at least two years post-surgery.
  Interventions: Drug: Encorafenib Pill; Drug: Binimetinib Pill
- Encorafenib and Binimetinib after Pathologic Complete Response (Experimental): Participants will receive 24 weeks of neoadjuvant encorafenib and binimetinib and then proceed to planned resection. If participants have pathologic complete response they will continue to receive encorafenib and binimetinib for 24 more weeks. Imaging will be conducted every 12 weeks for at least one year after surgery, and every 24 weeks for at least two years post-surgery.
  Interventions: Drug: Encorafenib Pill; Drug: Binimetinib Pill
- Encorafenib and Binimetinib after Non-Pathologic Complete Response (Experimental): Participants will receive 24 weeks of neoadjuvant encorafenib and binimetinib and then proceed to planned resection. If participants have non-pathologic complete response they will continue to receive encorafenib and binimetinib for 24 more weeks. Imaging will be conducted every 12 weeks for at least one year after surgery, and every 24 weeks for at least two years post-surgery.
  Interventions: Drug: Encorafenib Pill; Drug: Binimetinib Pill
- Nivolumab after Non-Pathologic Complete Response (Experimental): Participants will receive 24 weeks of neoadjuvant encorafenib and binimetinib and then proceed to planned resection. If participants have non-pathologic complete response they will receive nivolumab for 24 weeks. Imaging will be conducted every 12 weeks for at least one year after surgery, and every 24 weeks for at least two years post-surgery.
  Interventions: Drug: Encorafenib Pill; Drug: Binimetinib Pill; Drug: Nivolumab

INTERVENTIONS:
Drug: Encorafenib Pill — Encorafenib 450 mg will be administered orally once per day in continuous 28-day cycles
Drug: Binimetinib Pill — Binimetinib 45 mg will be administered orally twice per day in continuous 28-day cycles
Drug: Nivolumab — Nivolumab will be administered at a dose of 480 mg IV infusion over 30 minutes every 4 weeks.
  Arms: Nivolumab after Non-Pathologic Complete Response

SUMMARY:
The purpose of this study is to assess rate of disease relapse and hazard rate of disease relapse after neoadjuvant therapy based on the statuses of pathologic complete response or non-pathologic complete response, and postoperative adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of informed consent
* Histologically confirmed diagnosis of melanoma. Any primary or unknown origin is permitted.
* Melanoma must have a BRAFV600 mutation (using a CLIA-validated assay), either stage III (B/C/D) or Stage IV (AJCC 8th edition).
* ECOG performance status ≤ 2
* Adequate laboratory parameters as well:
* a. Hemoglobin ≥ 8 g/dL.
* b. Platelets ≥ 75 × 109/L;
* c. AST and ALT ≤ 2.5 × ULN; in participants with liver metastases ≤ 5 × ULN;
* d. Total bilirubin ≤ 1.5 × ULN and < 2 mg/dL; OR total bilirubin >1.5 × ULN with indirect bilirubin < 1.5 × ULN;
* e. Serum creatinine ≤ 2.0 × ULN
* Female participants of childbearing potential as described in protocol, must have a negative serum or urine β-HCG test result. Female participants of childbearing potential must agree to use methods of contraception that are highly effective or acceptable, as described in Section 4.3.1. Participants must agree to not use hormonal contraceptives, as encorafenib can result in decreased concentration and loss of efficacy. Male participants must agree to use methods of contraception that are highly effective or acceptable per protocol.

Exclusion Criteria:

* Participants may have received prior therapy with BRAF and/or a MEK inhibitor if it was completed at least 6 months prior to study enrollment. Patients who had prior disease progression while on BRAF/MEK inhibitor therapy are not eligible. (Progression after stopping treatment is permitted.) Participants may have received prior therapy an anti-PD-1/PD-L1 or CTLA-4 inhibitor.
* Participants must not have had adverse events related to encorafenib and/or binimetinib specifically, that required discontinuation of one or both drugs due to toxicity.
* Participants who have had major surgery or radiotherapy ≤ 14 days prior to start of study treatment or who have not recovered from side effects of such procedure.
* Participants must be willing to avoid consuming grapefruit, pomegranates, star fruits, Seville oranges or products containing the juice during the study while they are taking encorafenib/binimetinib.
* Uncontrolled or symptomatic brain metastases or leptomeningeal carcinomatosis that are not stable, require steroids, are potentially life-threatening or have required radiation within 28 days prior to starting study drug. Patients with previously treated brain metastases may participate provided they are stable (e.g.,without evidence of progression by radiographic imaging for at least 28 days before the first dose of study treatment and neurologic symptoms have returned to baseline).
* Impaired cardiovascular function as below:
* a. Congestive heart failure requiring treatment (New York Heart Association Grade ≥ 3);
* b. presence of uncontrolled atrial fibrillation or uncontrolled paroxysmal supraventricular tachycardia
* c. Baseline QTcF interval ≥ 500 ms.
* Known history of retinal vein occlusion (RVO)
* Current use of a prohibited medication (including herbal medications, supplements, or foods), as described in protocol, or use of a prohibited medication ≤ 1 week prior to the start of study treatment.
* Participants with a prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Participants with known human immunodeficiency virus (HIV)-infection are eligible providing they are on effective anti-retroviral therapy and have undetectable viral load at their most recent viral load test and within 90 days prior to randomization.
* Participants with a known history of hepatitis C virus (HCV) infection must have been treated and cured. Participants with HCV infection who are currently on treatment must have an undetectable HCV viral load prior to randomization.
* Pregnancy or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-05-24 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Rate of Disease Relapse | After surgery up to 24 weeks
  Investigators will estimate the rate of disease relapse after neoadjuvant therapy based on pathologic complete response status and postoperative adjuvant therapy within each arm.

SECONDARY OUTCOMES:
Relapse Free Survival | After surgery up to 24 weeks
  Relapse free survival is defined as time from surgery until disease relapse
Rate of Pathologic Complete Response | At 26 weeks
  Investigators will measure the rate of pathologic complete response after surgery.
Rate of Non-Pathologic Complete Response | At 26 weeks
  Investigators will measure the rate of non-pathologic complete response after surgery.
Overall Response Rate | Up to 26 weeks
  Overall response rate will be measured after neoadjuvant therapy (for participants who have measurable disease per RECIST 1.1 at start of neoadjuvant therapy).
Overall Survival | After surgery, up to 5 years
  Overall survival will be measured from time of surgery to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Eroglu, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States